CLINICAL TRIAL: NCT06865300
Title: Effects of Pretreatment with Different Doses of Lidocaine on Injection Pain and Rocuronium-induced Withdrawal Response
Brief Title: Effects of Pretreatment with Different Doses of Lidocaine on Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Azime Bulut, Associate Professor in the Department of Anesthesiology and Reanimation, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Mücahit
Record Dates: First submitted 2025-02-09; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Rocuronium Adverse Reaction; Lidocaine Adverse Reaction
Keywords: rocuronium; lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Injection of serum physiologic that contains no drug. (Placebo Comparator): We injected serum physiologic that contains no drug before injection of rocuronium and recorded pain score.
  Interventions: Drug: serum physiologic
- 40 mg lidocain group (Experimental): We injected 40 mg lidocain for the prevention of injection pain caused by rocuronium. We injected 0.06 mg/kg rocurunium and recorded pain by using visual analog scale.
  Interventions: Drug: Lidocain 40 mg
- 1 mg/kg lidocain group (Experimental): We injected 1 mg/kg lidocain for the prevention of injection pain caused by rocuronium. We injected 0.06 mg/kg rocurunium and recorded pain score by using visual analog scale.
  Interventions: Drug: lidocain 1 mg/kg

INTERVENTIONS:
Drug: Lidocain 40 mg — We injected 40 mg lidocain before rocuronium injection. Then we recorded pain score by using visual analog scale.
  Other Names: Lidocain; 40 mg lidocain
  Arms: 40 mg lidocain group
Drug: lidocain 1 mg/kg — We injected 1 mg/kg lidocain before rocuronium injection. Then we recorded pain score by using visual analog scale.
  Other Names: lidocain; 1 mg/kg lidocain
  Arms: 1 mg/kg lidocain group
Drug: serum physiologic — We injected serum physiologic before rocuronium injection. Then we recorded pain score by using visual analog scale.
  Other Names: izotonic fluid
  Arms: Injection of serum physiologic that contains no drug.

SUMMARY:
One of the medications administered to patients in general anesthesia practice is rocuronium, which causes pain during intravenous administration. It is known that a drug containing lidocaine as the active ingredient can reduce the pain caused by rocuronium in different doses. The effective dose of lidocaine remains a topic of debate. In our study, we aimed to investigate the efficacy of two different doses of lidocaine. No adverse effects are expected from this medication.

DETAILED DESCRIPTION:
The patients were randomly divided into three groups by a simple drawing-lots method: control group (Group C), 40 mg lidocaine group (Group L) and 1 mg/kg lidocaine group (Group L1). All patients were taken to the operating room without premedication and standard monitoring was applied. A 20 G intravenous catheter was inserted on the dorsum of the patients' non-dominant hand, and 100 ml/hour of physiological saline solution was infused over a 5-minute period. After randomization, 5 ml of isotonic solution was administered to the control group, 40 mg of lidocaine to the L group, and 1 mg kg-1 of lidocaine intravenously to the L1 group. Patients were administered 0.06 mg/kg of rocuronium, and they were asked, "Do you feel any pain or discomfort in your arm?" The pain intensity expressed by the patient was evaluated and recorded using the 5-point pain scale. After induction and intubation, the patients' blood pressure, pulse, and saturation values were recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged between 18 and 65 with ASA I and II

Exclusion Criteria:

* Chronic sedative anxiolytic use
* Those with ASA III and higher
* Patients under 18 and over 65 years of age
* Those with severe COPD, asthma, or reactive airway disease
* Patients with a history of neuropsychiatric or neurological diseases
* Those with infections on the back of the hand
* Pregnant women
* Patients who will undergo rapid induction
* Patients with liver and kidney dysfunction
* Those with a history of thrombophlebitis
* Patients with muscle diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Visual analog score after the injection | From enrollment to the end of injection at 5 minutes.
  We described Visual analog scale to the patient before the day of surgery. On the visual analog scale, a score of 10 is the worst pain in life, while a score of 0 is no pain. The patient is asked to give a score to his pain caused by rocuronium injection and the score is recorded.

SECONDARY OUTCOMES:
Changes on heart rate | Hemodynamic parameters were recorded 5 minutes intervals. Adverse effects of the drug were observed during 5 minutes after the injection.
  All patients who will receive general anesthesia are routinely monitored with electrocardiogram, noninvazive blood pressure and oxygen saturation. We recorded heart rate as beat per minute before and after the injections during 20 minutes.
Changes on noninvasive blood pressure | Hemodynamic parameters were recorded 5 minutes intervals. Adverse effects of the drug were observed during 5 minutes after the injection.
  All patients who will receive general anesthesia are routinely monitored with electrocardiogram, noninvazive blood pressure and oxygen saturation. We recorded noninvasive blood pressure as mmHg before and after the injections during 20 minutes.
Changes on oxygen saturation | Hemodynamic parameters were recorded 5 minutes intervals.
  All patients who will receive general anesthesia are routinely monitored with electrocardiogram, noninvazive blood pressure and oxygen saturation. We recorded oxygen saturation as percentage before and after the injections during 20 minutes.
Adverse effects | Adverse effects of the drug were observed during 5 minutes after the injection.
  After the injection of the drug we observed any side effect such as metallic taste, erythema, swelling, itching, allergic reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Azime Bulut, Study Director — Giresun University
Locations (2):
- Turkey (Türkiye) (2):
  - Giresun University, Giresun, Turkey
  - Giresun Training and Research Hospital, Giresun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh M, Chauhan H, Rath GP, Prabhakar H, Bithal PK, Dash HH. Effect of narcotic pretreatment on pain after rocuronium injection: a randomized, double-blind controlled comparison with lidocaine. J Anesth. 2007;21(4):510-2. doi: 10.1007/s00540-007-0560-8. Epub 2007 Nov 1. PMID 18008122
- [Background] Chiarella AB, Jolly DT, Huston CM, Clanachan AS. Comparison of four strategies to reduce the pain associated with intravenous administration of rocuronium. Br J Anaesth. 2003 Mar;90(3):377-9. doi: 10.1093/bja/aeg054. PMID 12594153
- [Background] Ergil J, Kavak Akelma F, Ozkan D, Bumin Aydin G, Gurel A, Akinci M. Effects of pretreatment with esmolol and lidocaine on injection pain and rocuronium-induced withdrawal response. Turk J Med Sci. 2015;45(4):959-63. doi: 10.3906/sag-1311-79. PMID 26422874
- [Background] Ahmad N, Choy CY, Aris EA, Balan S. Preventing the withdrawal response associated with rocuronium injection: a comparison of fentanyl with lidocaine. Anesth Analg. 2005 Apr;100(4):987-990. doi: 10.1213/01.ANE.0000147790.76114.3A. PMID 15781511
- [Background] Cheong KF, Wong WH. Pain on injection of rocuronium: influence of two doses of lidocaine pretreatment. Br J Anaesth. 2000 Jan;84(1):106-7. doi: 10.1093/oxfordjournals.bja.a013364. PMID 10740559